CLINICAL TRIAL: NCT02593890
Title: Breast Surgery Recovery: The Clinical and Psychosocial Impact of THEYA Recovery Range
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Claire Kelly (Industry)
Collaborators: University College Dublin (Other); Irish Research Council (Other)
Responsible Party: Sponsor-Investigator, Claire Kelly, Claire Kelly, Theya
Organization: Theya (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: THEYARCT2015
Record Dates: First submitted 2015-10-14; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Surgery; Mastectomy; Lumpectomy; Post-operative; Bra; Lingerie; Body Image; Psycho-social; Impact
MeSH Terms: conditions — Breast Neoplasms; Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Arm A: Participants will be fitted with the THEYA Recovery bra
  Interventions: Device: THEYA Recovery Range
- Control (No Intervention): Arm B: Participants will be recommended or fitted with current recommended bra used in each hospital by the Breast Care Nurse Specialist

INTERVENTIONS:
Device: THEYA Recovery Range — Post-operative Lingerie made from viscose derived bamboo
  Arms: Intervention

SUMMARY:
A randomised interventional comparative control study will be undertaken to compare the THEYA Recovery Range postoperatively for patients undergoing wider lumpectomies, partial mastectomies and total mastectomies to current practice using a mixed method combining quantitative and qualitative instruments. 100 female participants are hoped to be recruited following breast surgery after a newly diagnosed breast cancer.

This study will answer the research question:- "What is the clinical and psychosocial impact of the THEYA Recovery Range in comparison to recommended practice during and after breast cancer treatment?" This study will leverage the findings of a pilot study conducted by Applied Research Connected Healthcare (ARCH) measuring the usability of the THEYA Recovery Range.

This study aims to assess the participants' experience of recovery in the immediate post-operative period and the psychosocial effect of THEYA Recovery Range in comparison to current recommended practice.

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer worldwide, and the most frequent cancer among females with nearly 1.67 million new cases diagnosed in 2012 (WHO, 2012). Due to population increases, health service and cancer awareness, more women are diagnosed with breast cancer each year. Advances in diagnosis and in treatment have seen an increase in survival from breast cancer for Irish women in recent years (ABC, 2010). In Ireland, after non-melanoma skin cancer, breast cancer is the most common tumour diagnosed in women in 2008-2010. With an average annual amount of 2,767 women diagnosed with breast cancer in 2008-2010 (NCRI, 2013). As a result, more women are living with the permanent effects of breast cancer (Gho et al., 2010).

For patients' newly diagnosed with breast cancer, surgery is the first choice of treatment. 84% of females receive surgery as a form of treatment, be it as a single modality or in combination with radiotherapy, chemotherapy and/or hormone therapy (NCRI, 2012).

A randomized interventional comparative control study will be undertaken to compare the THEYA Recovery Range postoperatively for patients undergoing wider lumpectomies, partial mastectomies and total mastectomies using a mixed method combining quantitative and qualitative instruments. 100 female participants are hoped to be recruited following breast surgery after a newly diagnosed breast cancer.

Who can participate? Women over the age of 18 years with no upper age limit, with a newly diagnosed breast cancer that are planned to undergo breast surgery as treatment in a 3 month period from recruitment.

What does the study involve? Participants will be randomly assigned, by use of a sealed envelope into two groups: an intervention and a control group.

Women in the intervention group will be fitted by the investigator with a THEYA Recovery bra.

Women in the control group will have standard post-operative care, with recommended bra or fitted by the Breast Care Nurse Specialist.

All participants will complete three questionnaires before fitting : The Breast Q, The Body Image Scale and the EQ 5D 3L.

All participants will be asked to continue wearing bra for a period of three to four weeks, then re-assessed on return visit, with re-assessment of the three questionnaires. 30 partcipants will be randomly selected from the sealed envelope to undergo a semi-structured interview, in order to gain a better understanding of their experience.

What are the possible benefits and risks of participating? The benefits for participating include receiving the same level of care, and for those undergoing lumpectomy a free bra. The study aims to evaluate the patients requirements in post-operative lingerie in order to help and further assiss these women. As this is an area of minimal research. There are no risks envisaged from participating in this study.

Where is the study run from? The study is ran from The Beacon Hospital, Mater Misericordiae University Hospital, Mater Private Hospital and St.James's Hospital.

When is the study starting and how long is it expected to run for? The study is planned to start in November 2015 and is expected to run until December 2016.

Who is funding the study? The study is being funded from the Irish Research Council and THEYA as part of an Employment Based PostGraduate Award.

Who is the main contact? Claire Kelly, Researcher.

claire@theya.healthcare

ELIGIBILITY:
Inclusion Criteria:

1. Female over the age of 18 years, with no maximum age limit once all other criteria are met.
2. Have a comprehensive understanding and fluency of the English language with the ability to provide informed consent.
3. Be scheduled to undergo a mastectomy or lumpectomy for a new first time diagnosis of breast cancer within a 3 month period of recruitment - as this cohort are the principal users of post-surgery bras.
4. No pre-existing severe co-morbidities and / or documented psychological diagnosis i.e. depression, severe chronic disease - as we do not want to over-burden a person who has any ailments other than their surgery discomfort. As well as that, the bra is designed to help recovery from breast surgery, and having further ailments may alter data we receive.
5. Be available for the full duration of the study which will be 3 months from recruitment to post-assessment.

Exclusion Criteria:

1. Are under the age of 18 years.
2. Do not have intellectual capacity to provide informed consent.
3. Are not scheduled to undergo a mastectomy or lumpectomy within a 3 month period of recruitment.
4. Have pre-existing severe co-morbiditie(s) and / or documented psychological diagnosis, as the diagnosis of breast cancer is challenging enough and it may exacerbate any psychological condition, and the researcher would like to avoid any perceived additional stress for them.
5. Those that are not fluent English speakers, grossly hearing or speech impaired.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
THEYA Recovery post-surgery bra impacted on the participant's quality of life using the 2009 EuroQol Group questionnaire EQ-5D-5L. | Four weeks
  The EQ-5D-3L measures the respondent's health related Quality of Life
  100 represents the "Best imaginable health status' and 0 represents the 'Worst imaginable health status'

SECONDARY OUTCOMES:
THEYA Recovery post-surgery bra impact on Body Image using The Body Image Scale (Hopwood et al, 2001) | Four weeks
  The scale consists of ten questions for assessment. Response options range from ''not at all'' (score 0), ''a little'' (score 1), ''quite a bit'' (score 2) to ''very much'' (score 3).
  A total score ranging from 0 to 30 per patient with 0 representing no distress or symptoms, whereas increasing scores represent increasing distress and symptoms.
THEYA Recovery post-surgery bra impact on feminity, sexuality, pain, sleep distrubance, body image assessed by The Breast Q Mastectomy or The Breast Q Breast Conserving Treatment, derived by Memorial Sloan Kettering. | Four weeks
  Breast-Q Questionnaire (measure through questionnaires the quality of life and psychosocial indicators specific to breast cancer survivors)

OTHER OUTCOMES:
The participants' explained perceptions of the comfort, functionality and reported levels of health and wellbeing compared to the control, following a semi-structured interview. Measured through qualitative analysis using NVivo package. | Four weeks
  A qualitative semi-structured interview designed by the researcher to evaluate the lived experience of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda McCann, PhD, Study Director — University College Dublin